CLINICAL TRIAL: NCT01175317
Title: Does Hemodynamic Optimization During and After Colorectal Surgery Result in Improved Intestinal Perfusion, Sustained Intestinal Barrier and Improved Postoperative Recovery?
Brief Title: Improvement of Fluid Balance in Patients Undergoing Surgery of the Colon and Rectum
Acronym: HOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 09-2-089
Record Dates: First submitted 2010-07-29; First posted 2010-08-04 (Estimated); Results first posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Carcinoma
Keywords: Hemodynamic optimization; Enhanced recovery after surgery; Goal-directed fluid
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goal-directed fluid optimization (Experimental): Fluid administration and optimization based on cardiac output findings during surgery and during the first 8 hours of the postoperative phase.
  Interventions: Procedure: Goal-directed fluid optimization
- Regimen based on expertise anaesthesist (Other): Fluid regimen based on expertise anaesthesist
  Interventions: Other: Regimen based on expertise anaesthesist

INTERVENTIONS:
Procedure: Goal-directed fluid optimization — Fluid administration and optimization based on cardiac output findings during surgery and during the first 8 hours of the postoperative phase.
  Arms: Goal-directed fluid optimization
Other: Regimen based on expertise anaesthesist — Fluid regimen based on expertise anaesthesist
  Arms: Regimen based on expertise anaesthesist

SUMMARY:
58 patients undergoing surgery of the large bowel are divided into two groups. The control group will receive standard care. The intervention group will receive standard care plus optimization of the blood circulation based on in- or decrease of the output of the heart. Between group differences are measured primarily by markers of intestinal damage in plasma and urine. Also CO2 pressure in the stomach lumen is measured (reflecting blood supply to the gut).

The investigators hypothesize that the intervention group will have less intestinal damage, improved blood supply to the bowel and improved recovery of the operation compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective colorectal surgery with anastomosis;
* Minimum age 18 years;
* Giving informed consent.

Exclusion Criteria:

* Other causes of intestinal damage: eg. IBD, occlusive disease;
* Steroid use;
* Esophageal varices and other esophageal disease;
* Aortic valve disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten F Von Meyenfeldt, MD, PhD, Study Director — Maastricht University Medical Center; Martijn Poeze, MD, PhD, Study Director — Maastricht University Medical Center; Geerard L Beets, MD, PhD, Study Director — Maastricht University Hospital; Wim A Buurman, PhD, Study Director — Maastricht University
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion period: july 2010 - october 2013 at single University Hospital: Maastricht University Medical Center.
Pre-assignment Details: Patient inclusion rate was lower than expected. Main reason was unwillingness to participate, as extra nasal probes would remain in situ after surgery.
Period: Overall Study
Arm/Group | Goal-directed Fluid Optimization | Regimen Based on Expertise Anaesthesist
Started | 27 | 31
Completed | 27 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Goald-directed Fluid Optimization: Fluid administration and optimization based on cardiac output findings during surgery and during the first 8 hours of the postoperative phase.
- Total: Total of all reporting groups
Arm/Group | Goald-directed Fluid Optimization | Regimen Based on Expertise Anaesthesist | Total
Number analyzed (Participants) | 27 | 31 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 13 | 22
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (10.8) | 67.6 (10.0) | 68.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 21 | 20 | 41
Region of Enrollment [Number; unit: participants]
  Netherlands | 27 | 31 | 58

OUTCOME MEASURES:

1. Primary Outcome: Peak Value of I-FABP
Description: Intestinal-Fatty Acid Binding Protein (a marker of intestinal damage) is measured in plasma.
  The primary outcome measure is the difference in peak values of I-FABP between the control group and the intervention group.
Time Frame: 1 hour postoperatively
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Goal-directed Fluid Optimization | Regimen Based on Expertise Anaesthesist
Number analyzed (Participants) | 27 | 31
pg/mL | 440.8 (251.6) | 522.4 (759.9)

2. Secondary Outcome: Average Intraoperative CO2 Gap
Description: The CO2 gap (difference arterial pCO2 and pCO2 of the stomach lumen) reflects global intestinal perfusion status and is measured every 15 minutes intraoperatively and every 60 minutes during the first 8 hours postoperatively.
  Intraoperative measurements were averaged per individual patient, producing the average intraoperative CO2 gap.
Time Frame: Average intraoperative CO2 gap
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Goal-directed Fluid Optimization | Regimen Based on Expertise Anaesthesist
Number analyzed (Participants) | 27 | 31
kPa | -0.1 (0.6) | 0.4 (0.5)

ADVERSE EVENTS:
Arm/Group | Goal-directed Fluid Optimization | Regimen Based on Expertise Anaesthesist
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/31

LIMITATIONS AND CAVEATS:
Tolerance of esophageal Doppler probe postoperatively was low. Therefore, optimization based on cardiac output could only be achieved within 3 hours in most patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes